CLINICAL TRIAL: NCT05502211
Title: A Comparison Between Ketamine-lidocaine Versus Ketamine-fentanyl for Induction on the Hemodynamic Effects in Patients With Coronary Artery Disease and Left Ventricular Systolic Dysfunction :( A Randomized Controlled Study
Brief Title: A Comparison Between Ketamine-lidocaine Versus Ketamine-fentanyl for Induction on the Hemodynamic Effects in Patients With Coronary Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ayman Abougabal, Dr Abougabal, Kasr El Aini Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: MS-230-2022
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Induction of General Anesthesia
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Experimental)
  Interventions: Drug: Lidocaine IV
- Fentanyl (Active Comparator)
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — induction of anaesthesia using fentanyl
  Arms: Fentanyl
Drug: Lidocaine IV — induction of anesthesia using lidocaine
  Arms: Lidocaine

SUMMARY:
Patients with coronary artery disease (CAD) and left ventricular systolic dysfunction (LVSD) presenting for coronary artery bypass grafting (CABG) represent a high-risk group among the cardiac surgical population. Anesthetic management of these patients is challenging due to increased risk of perioperative hypotension and subsequently increased risk of postoperative morbidity and mortality. Post induction hypotension is a modifiable risk that can be largely prevented by adjusting the technique for anesthesia induction. There is no consensus on the use of certain anesthetic induction techniques for patients CAD and left ventricular dysfunction. Anesthesia induction techniques for cardiovascular surgery are usually based on considerations such as hemodynamic stability, effects on myocardial oxygen supply, and demand and minimizing intubation stress response.To the best of our knowledge, there is no previous data comparing the efficacy of adding lidocaine versus fentanyl to the induction of anesthesia with ketamine in patients with poor ventricular function.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be patients with coronary artery disease and moderate to severe left ventricular dysfunction (ejection fraction < 40%), ASA physical status II-IV that will be scheduled for elective CABG surgery.

Exclusion Criteria:

* Patients with associated valvular heart disease, persistent arrhythmias, congestive cardiac failure, on mechanical ventilation, intra-aortic balloon pump (IABP), emergency surgery, and those with known allergy to any of the study's drugs, severe systemic non-cardiac disease; will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
incidence of hypotension | 15 minutes post inductin
  the number of patients who will develop hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Abougabal, MD, Study Chair — lecturer of anesthesia Kasr Al Ainy hospital
Locations (2):
- Egypt (2):
  - Kasr Al Ainy, Cairo
  - Kasr al ainy, Cairo

IPD SHARING:
Plan to Share IPD: No